CLINICAL TRIAL: NCT03732651
Title: The Impact of Non-pulsatile Perfusion on Cerebral Blood Flow and Brain Oxygenation
Brief Title: The Impact of Non-pulsatile Blood Flow on CO2-Reactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Cecilia Veraar, Cecilia Veraar, Medical University of Vienna
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1018730
Record Dates: First submitted 2018-10-30; First posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Cerebrovascular Circulation

STUDY DESIGN:
Intervention Model Description: Each patient served as his own control.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-pulsatile blood flow (Experimental)
  Interventions: Procedure: alteration of PaCO2 level
- pulsatile blood flow (Experimental)
  Interventions: Procedure: alteration of PaCO2 level

INTERVENTIONS:
Procedure: alteration of PaCO2 level — step changes between 30, 40 and 50 mmHg

SUMMARY:
The investigators hypothezised that CO2-reactivity of cerebral vessels is affected by systemic non-pulsatile blood flow. Patients undergoing elective cardiac surgery with CPB were enrolled in this prospective case control study. Blood flow velocity in the middle cerebral artery as well as regional cerebral oxygenation was determined during step changes of PaCO2 between 30, 40, and 50 mmHg. Measurements were conducted intraoperatively during non-pulsatile as well as postoperatively after admission to the ICU under pulsatile blood flow.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* Carotid artery stenosis (> 50%)
* Neurological pathologies
* COPD with CO2 retention
* Women of childbearing age

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-06-11 (Actual); Primary Completion 2012-10-11 (Actual); Study Completion 2013-12-02 (Actual)

PRIMARY OUTCOMES:
CO2- Reactivity of cerebral vessels during cardiopulmonary bypass using nonpulsatile blood flow and postoperative on ICU under physiological pulsatile blood flow | first time-point: intraoperative, during cardiopulmonary bypass, duration up to 300minutes. Second time-point: on ICU, postoperatively under pulsatile blood flow, duration of measurement up to 100minutes for each patient
  Relation between PaCO2 level and cerebral blood flow velocity will be assessed during non-pulsatile and pulsatile blood flow. Measurements will be performed using trancranial doppler to measure flow velocity of the middle cerebral artery. Further, NIRS will be used to measure oxygen saturation of the brain. Measurements will be performed during step changes of PaCO2 (at 30mmHg, 40mmHg and 50mmHg.

CONTACTS AND LOCATIONS:
Locations (1):
- medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Veraar CM, Rinosl H, Kuhn K, Skhirtladze-Dworschak K, Felli A, Mouhieddine M, Menger J, Pataraia E, Ankersmit HJ, Dworschak M. Non-pulsatile blood flow is associated with enhanced cerebrovascular carbon dioxide reactivity and an attenuated relationship between cerebral blood flow and regional brain oxygenation. Crit Care. 2019 Dec 30;23(1):426. doi: 10.1186/s13054-019-2671-7. PMID 31888721